CLINICAL TRIAL: NCT00582361
Title: Vacuum Assisted Closure as a Treatment for Open Fractures
Acronym: VAC-OF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F010316004
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2012-05

CONDITIONS: Orthopaedic Traumatic Open Fractures
Keywords: Open Fractures; Vacuum Assisted Closure (VAC) device; Irrigation and Debridement
MeSH Terms: conditions — Fractures, Open | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1, A (Active Comparator): Group A patients will have a standard dressing applied following initial treatment of their open fracture.
  Interventions: Procedure: Standard Wound Dressing
- 2, B (Experimental): Group B patients will have a Vacuum Assisted Closure (VAC) device applied following initial treatment of their open fracture.
  Interventions: Device: VAC

INTERVENTIONS:
Procedure: Standard Wound Dressing — Group A patients will have a standard dressing applied following initial treatment of their open fracture. They will return to the operating room approximately 48 hours following the initial trauma, and approximately every 48 hours thereafter, for irrigation and debridement and concomitant wound cultures (qualitative and quantitative) until such time as the wound is judged by the surgeon to be ready for either delayed primary closure or flap/skin graft coverage.
  Arms: 1, A
Device: VAC — Group B patients will have a Vacuum Assisted Closure (VAC) device applied following initial treatment of their open fracture. They will return to the operating room approximately 48 hours following the initial trauma, and approximately every 48 hours thereafter, for irrigation and debridement and concomitant wound cultures (qualitative and quantitative) until such time as the wound is judged by the surgeon to be ready for either delayed primary closure or flap/skin graft coverage.
  Other Names: Vacuum Assisted Closure (VAC)
  Arms: 2, B

SUMMARY:
This project is designed as a prospective, randomized, comparative study evaluating the use of a negative pressure vacuum device in treating traumatic wounds sustained associated with an open fracture.

DETAILED DESCRIPTION:
Soft tissue injury following an open fracture is a significant problem following surgical treatment of traumatic skeletal injuries. The soft tissue injury results from a combination of the initiating trauma and additional tissue injury during surgery. Current treatment includes open reduction and internal fixation versus external fixation, irrigation and debridement following admission, decreased activity (non weight bearing status on the injured extremity), maintaining the patient as an inpatient in the hospital, repeated irrigation and debridements (36-72 hours following the initial trauma) with concomitant wound culturing until which time it is determined that either delayed primary closure, or skin grafting with/without flap coverage should be attempted.

All patients in the study will be treated with the appropriate empiric antibiotic regimen until wound culture results justify modification for antibiotic sensitivity/resistance reasons. In general, barring patient allergy, the empiric antibiotic regimen will adhere to the Gustilo and Anderson classification as follows:

Grade I : Ancef Grade II : Ancef and Gentamicin or Zosyn Grade III : Ancef, Gentamicin or Zosyn, and add a Penicillin for grade IIIB open fractures.

All wounds will be assessed initially at admission following the Gustilo and Anderson classification for open fractures. Subsequent wound assessments in the operating room will be graded according to the following descriptive scale:

Type A wound: Abundant granulation tissue, ready for closure. Type B Wound: Granulation tissue present but inadequate for closure, Wound is clinically clean appearing. Type C Wound: No granulation tissue, no gross purulence. Type D Wound: Gross purulence/infected wound, no granulation tissue.

The outcome variables consist of the intraoperative and postoperative adverse device effects recorded in the medical record and on the study data collection form, time to wound closure, intraoperative and postoperative complications recorded in medical record and on the study data collection form. Clinical photographs of the wounds will be taken with a digital camera at the time of admission to the study, and during each subsequent trip to the operating room (every 48-72 hours). We will also record the injury severity score for all multiple trauma patients recorded at the time of injury in the medical record and on the study data collection form, and soft tissue score according to Gustillo and Anderson for open injuries in the medical record and on the study data collection form. Baseline serum albumin and total lymphocyte counts will be taken on admission to evaluate baseline nutritional and immunologic status at the time of injury. All patients in the Intensive Care Units will have daily weights, fluid balances, and nutritional intake documented. Resuscitation data will also be recorded from the trauma room, including fluids, blood, and base deficit. The effects will be measured by clinical examination and will be augmented with culture data for any wounds that require surgical intervention.

Patients who have an open fracture and who give informed consent to enter the study will be randomized into two groups. Group A will be patients treated with a return to the operating room approximately 48 hours following the initial trauma, and approximately every 48 hours thereafter, for irrigation and debridement and concomitant wound cultures (qualitative and quantitative) until which time the wound is judged by the surgeon to be ready for either delayed primary closure or flap/skin graft coverage. Group B will be patients treated with a VAC negative pressure device following the initial surgical irrigation and debridement. Group B patients will return to the operating room approximately 48 hours following the initial irrigation and debridement for VAC removal, wound cultures (qualitative and quantitative), repeat irrigation and debridement, and wound evaluation by the surgeon for possible delayed closure versus reapplication of the VAC device. Group B patients will also be returned to the operating room approximately every 48 hours thereafter for irrigation and debridement and concomitant wound cultures (qualitative and quantitative) until the wound is judged ready for coverage or closure by the surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has sustained an open fracture that requires surgical irrigation and debridement.
* No gross clinical evidence of infection.

Exclusion Criteria:

* A grossly infected open wound. Infection will be defined by clinical signs and symptoms of infection that include increasing drainage, increasing pain, purulent drainage, and increasing erythema. Any wounds that are thought to be infected will be cultured to confirm the diagnosis.
* A surgical incision that can not be covered with VAC sponges and a water impermeable sheet (such as Ioban or Tegaderm) to achieve a closed vacuum environment over the wound.
* Wounds associated with the surgical incision that are intentionally left open to heal with either a delayed primary closure or secondary granulation
* Abnormal coagulation leading to an expanding hematoma that will require surgical debridement.
* Pregnant women.
* Inability or unwillingness to comply with protocol.
* Patients or family members who are unable or unwilling to sign study informed consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2001-06; Primary Completion 2008-09 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rena L Stewart, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Orthopaedic Trauma, Birmingham, Alabama, United States

REFERENCES:
- [Background] Parrett BM, Matros E, Pribaz JJ, Orgill DP. Lower extremity trauma: trends in the management of soft-tissue reconstruction of open tibia-fibula fractures. Plast Reconstr Surg. 2006 Apr;117(4):1315-22; discussion 1323-4. doi: 10.1097/01.prs.0000204959.18136.36. PMID 16582806
- [Background] Steiert AE, Partenheimer A, Schreiber T, Muehlberger T, Krettek C, Lahoda LU, Vogt PM. [The V.A.C. system (vacuum assisted closure) as bridging between primary osteosynthesis in conjunction with functional reconstructed of soft tissue--open fractures type 2 and type 3]. Zentralbl Chir. 2004 May;129 Suppl 1:S98-100. doi: 10.1055/s-2004-822658. German. PMID 15168301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients admitted through the emergency department that met the criteria for the study were approached.
Groups:
- Standard Dressing Group (1, A): Group 1,A subjects will have a standard dressing applied following initial treatment of their open fracture.
- Vacuum Assisted Closure Group (2, B): Group 2,B subjects will have a Vacuum Assisted Closure (VAC) device applied following initial treatment of their open fracture.
Period: Overall Study
Arm/Group | Standard Dressing Group (1, A) | Vacuum Assisted Closure Group (2, B)
Started | 25 | 38
Completed | 25 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dressing Group (1, A) | Vacuum Assisted Closure Group (2, B) | Total
Number analyzed (Participants) | 25 | 38 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 35 | 58
  >=65 years | 2 | 3 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (16) | 38 (15) | 41 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 15 | 28 | 43
Region of Enrollment [Number; unit: participants]
  United States | 25 | 38 | 63

OUTCOME MEASURES:

1. Primary Outcome: Healing of Orthopaedic Trauma Open Fractures
Description: Healing of the open wound following orthopaedic trauma open fracture surgery was measured in days. (The wound has healed adequately to permit closure)
Time Frame: from surgery to wound closure
Measure: Mean (Full Range); unit: use days
Arm/Group | Standard Dressing Group (1, A) | Vacuum Assisted Closure Group (2, B)
Number analyzed (Participants) | 23 | 35
use days | 3.2 [2 to 9] | 4.0 [2 to 11]

2. Primary Outcome: Infections
Description: Number of acute, delayed and deep wound infections.
Time Frame: Up to 12 months
Measure: Number; unit: Number of infections
Arm/Group | Standard Dressing Group (1, A) | Vacuum Assisted Closure Group (2, B)
Number analyzed (Participants) | 25 | 37
Number of infections | 7 | 2

ADVERSE EVENTS:
Time Frame: Through 12 months (date of surgery through 12 months)
Arm/Group | Standard Dressing Group (1, A) | Vacuum Assisted Closure Group (2, B)
Serious Adverse Events (participants affected / at risk) | 1/25 | 4/38
Other Adverse Events (participants affected / at risk) | 0/25 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dressing Group (1, A) (N=25) | Vacuum Assisted Closure Group (2, B) (N=38)
Nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Required Flap Coverage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Amputation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
None Noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No